CLINICAL TRIAL: NCT07145749
Title: Investigation of the Effects of Transtheoretical Theory-based Education Given to Individuals Followed in Amatem on Their Sexual Risk Taking, AIDS Knowledge Levels and Protection Self-efficacy: a Randomized Controlled Trial.
Brief Title: Examining the Effects of Theory-based Education on Individuals' Sexual Behavior.
Acronym: SEXUALRISK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Hülya İncirkuş Küçük, PhD Student, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: E-71522473-050.04-372987-197
Record Dates: First submitted 2024-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections; Sexual Behavior
MeSH Terms: conditions — HIV Infections; Sexual Behavior

STUDY DESIGN:
Intervention Model Description: The experimental group will receive 8 weeks of transtheoretical theory-based training and will be given a training booklet at the end of the training.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Since the training will be given to the experimental group in our study, it was not possible to provide double-blind researcher blindness in terms of blinding and masking. However, masking was applied wherever possible from the delivery of evaluations to the scoring and the initial assignment of individuals. The researcher who conducted the survey, made the random assignment, the researcher who made the statistical evaluation and the AMATEM personnel who drew the envelopes were blinded to the study. At the same time, the coded answer sheets will only be entered into the analysis program after the study is completed. Single-blind randomization will be provided by ensuring that the person who does the analysis does not know which individual the survey forms belong to. It was planned in a way that the experimental group would not meet the control group before and after the training program. In this way, cross-contamination of the experimental and control groups was prevented.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Transtheoretical theory-based education will be provided to individuals with substance use disorders face-to-face in 8 modes and each lesson will last 45 minutes. Weekly education stages of transtheoretical theory-based education: Week 1; Stage 1 (not thinking); Weeks 2 and 3, Stage 2 (Thinking/Intention); Weeks 4 and 5, Stage 3 (Preparation); Weeks 6 and 7, Stage 4 (taking action); Week 8, Stage 5 (Maintenance/Continuing).
  Interventions: Behavioral: Transtheoretical theory-based education; Other: Pre-test-after-test-re-test
- Control group (Other): No additional intervention will be applied.
  Interventions: Other: Pre-test-after-test-re-test

INTERVENTIONS:
Behavioral: Transtheoretical theory-based education — Transtheoretical theory-based education will be provided to individuals with substance use disorders face-to-face in 8 modes and each lesson will last 45 minutes. Weekly education stages of transtheoretical theory-based education: Week 1; Stage 1 (not thinking); Weeks 2 and 3, Stage 2 (Thinking/Intention); Weeks 4 and 5, Stage 3 (Preparation); Weeks 6 and 7, Stage 4 (taking action); Week 8, Stage 5 (Maintenance/Continuing).
  Arms: Experimental group
Other: Pre-test-after-test-re-test — Information Form, Sexual Risk Taking Scale, AIDS Knowledge Scale and AIDS Prevention Self-Efficacy Scale

SUMMARY:
The research was planned to examine the effect of the transtheoretic theory-based education given to individuals followed in AMATEM on their sexual risk-taking status, AIDS knowledge level and AIDS prevention self-efficacy.

Research Hypotheses H0: Transtheoretical theory-based education given to individuals followed in AMATEM has no effect on their sexual risk taking, AIDS knowledge level and protection self-efficacy.

H1-1: Transtheoretic theory-based education given to individuals followed in AMATEM has an effect on the level of sexual risk taking.

H1-2: The transtheoretic theory-based education given to individuals followed in AMATEM is A

DETAILED DESCRIPTION:
Substance abuse is a public health problem as old as human history. Globally, increasing substance use disorder has become a public health problem that harms individuals and then societies, and has negative effects on many dimensions such as economic, social and security. In addition to its history dating back to ancient times, the content and effects of the substances used have changed over time and spread more rapidly in societies as a result of the production of easily accessible concentrated forms. Substances of abuse are categorized in two ways. These include a variety of illegal and legally sanctioned substances. The most common types of illegal substances include cannabis, amphetamine, ketamine, methamphetamine, cocaine, ecstasy and heroin, which are largely banned in most countries. Tobacco and alcohol are two types of legally sanctioned substances that are widely used by different social groups across different societies and cultures. In the treatment of substance use disorder, behavioral change can be achieved with theory-based training provided in addition to pharmacological treatment. The theory-based approach in nursing practices increases the quality of health services provided and guides nurses. The Transtheoretical Model (TTM) or Stages of Change Model developed by Prochaska and Diclemente (1982) describes the change of healthy life behaviors in individuals in stages. As a result of the literature review, it was seen that the transtheoretical model is frequently used in order to reduce symptoms in addiction and other chronic diseases, improve health, and provide healthy life behaviors to individuals. The individuals followed in AMATEM, which constitute the sample of our research, are at greater risk of sexually transmitted HIV by exhibiting risky sexual behavior. It is thought that TTM-based training integrated into substance use treatment in order to reduce the tendency towards uncontrolled sexual behaviors as a result of substance use disorder and the risk of infectious diseases as a result will create healthy behavioral change in individuals.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate voluntarily in the study
* Age 18 years or older
* Under probation and receiving treatment at AMATEM
* Able to read and write (literate)

Exclusion Criteria:

* Presence of visual, hearing, or communication disorders
* Refusing to participate voluntarily in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Sexual Risk Taking Scale (SCRAS) | At the end of the planned training program (8 weeks); It will be applied as the final test. In order to measure the permanence of behavioral change after the training, the final test was planned to be repeated after an average of 2 months.
  It consists of a total of 10 items aimed at collecting information about risky sexual behaviors experienced by the person in the last 12 months and throughout his/her life. Five items of the scale are answered as yes-no, two items are answered as fill-in-the-blank, two items are answered as triple Likert type, and one item is answered as quadruple Likert type. The possible score from the scale is between 0 and 10, with higher scores indicating more sexual risk taking.The alpha internal consistency coefficient of the scale was found to be 0.71.
AIDS Knowledge Scale (AIS) | At the end of the planned training program (8 weeks); It will be applied as the final test. In order to measure the permanence of behavioral change after the training, the final test was planned to be repeated after an average of 2 months.
  The scale has 18 items. The total score varies between 0-18, with higher scores indicating more AIDS knowledge. The content validity index of the scale was found to be 0.98. The internal consistency of the scale was found to be 0.85 and the test-retest reliability was found to be 0.80.
AIDS Prevention Self-Efficacy Scale (AIPS) | At the end of the planned training program (8 weeks); It will be applied as the final test. In order to measure the permanence of behavioral change after the training, the final test was planned to be repeated after an average of 2 months.
  It is a five-point Likert-type scale with a total of 27 items. Scores on the scale range from 27 to 135, with higher scores indicating higher self-efficacy. The internal consistency coefficient of the total scale was found to be 0.93, and the test-retest reliability was found to be 0.85.

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya Sağlik Bilimleri Enstitüsü, Sakarya, Serdi̇van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin H, Liu Y, Zhang H, Zhu Z, Zhang X, Chang C. Assessment of a Text Message-Based Smoking Cessation Intervention for Adult Smokers in China: A Randomized Clinical Trial. JAMA Netw Open. 2023 Mar 1;6(3):e230301. doi: 10.1001/jamanetworkopen.2023.0301. PMID 36857056
- [Result] Leandro TA, Nunes MM, Teixeira IX, Lopes MVO, Araujo TL, Lima FET, Silva VMD. Development of middle-range theories in nursing. Rev Bras Enferm. 2020 Feb 10;73(1):e20170893. doi: 10.1590/0034-7167-2017-0893. eCollection 2020. English, Portuguese. PMID 32049218
- [Result] Evers YJ, Op den Camp KPL, Lenaers M, Dukers-Muijrers NHTM, Hoebe CJPA. Alcohol and drug use during sex and its association with sexually transmitted infections: a retrospective cohort study among young people aged under 25 years visiting Dutch STI clinics. Sex Transm Infect. 2023 Mar;99(2):97-103. doi: 10.1136/sextrans-2021-055355. Epub 2022 May 6. PMID 35523571
- [Result] Efrati Y, Kraus SW, Kaplan G. Common Features in Compulsive Sexual Behavior, Substance Use Disorders, Personality, Temperament, and Attachment-A Narrative Review. Int J Environ Res Public Health. 2021 Dec 28;19(1):296. doi: 10.3390/ijerph19010296. PMID 35010552
- [Result] Chun J. Public Health Threat of Tobacco and Substance Use in Asia: An Introduction to the Theme Issue. J Psychoactive Drugs. 2020 Jan-Mar;52(1):1-4. doi: 10.1080/02791072.2020.1717686. Epub 2020 Jan 22. PMID 31967534